CLINICAL TRIAL: NCT06451731
Title: Rehabilitation of Post-stroke Aphasia by a Single Protocol Targeting Phonological, Lexical, and Semantic Deficits With Speech Output Tasks: a Randomized Controlled Trial
Brief Title: Rehabilitation of Post-stroke Aphasia by Targeting Phonological, and Lexico-semantic Deficits With Speech Output Tasks
Acronym: PHOLEXSEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25C501
Record Dates: First submitted 2024-05-16; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Aphasia, Acquired; Stroke; Anomia
MeSH Terms: conditions — Aphasia; Stroke; Anomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHOLEXSEM (Experimental): Each session lasted 30 minutes, and comprised three sections, each lasting 10 minutes: Repetition, Semantic Feature Analysis (SFA), and Lexical retrieval.
  Repetition: 50 items for different kind of stimuli including: syllables, 2-syllable words and non-words; 2-syllable words and non-words with one consonant cluster; 3-syllable words and non-words; 3-syllable words and non-words with one consonant cluster, nuclear phrases.
  SFA: stimuli were 46 pictures of nouns, including living and non-living objects, controlled for frequency of use.
  Lexical retrieval phase: the patient was given three fluency tasks: a) 4 min of phonemic recall, b) 4 min of semantic recall, and c) 2 min of verb recall.
  Interventions: Behavioral: PHOLEXSEM
- PACE (Active Comparator): Three decks of cards - diversified by frequency of use - depicting nouns, were presented in sets of 4 cards each. In an exchange modality, the task consisted in understanding the noun chosen by the patient and, in turn, by the rehabilitator. Any communicative modality (oral, gestural, verbal, graphic) was allowed. Word difficulty was graded based on the frequency of use and semantic proximity or distance between target and distractors.
  Interventions: Behavioral: PACE

INTERVENTIONS:
Behavioral: PHOLEXSEM — Phonological, Lexical, and Semantic training
  Arms: PHOLEXSEM
Behavioral: PACE — See arm description
  Arms: PACE

SUMMARY:
Aphasia in brain-damaged adult patients refers "to the more or less complete loss of the ability to use language" resulting from acquired brain damage, typically of the left hemisphere. The defective spoken output of persons with aphasia (PWA) has anomia as a main clinical manifestation. Improving anomia is a main goal of any language treatment.

The present randomized controlled study assessed the effectiveness of a novel, two-week, rehabilitation protocol (PHOLEXSEM), focused on PHonological, SEmantic, and LExical deficits, aiming at improving lexical retrieval, and, generally, spoken output.

The effects of the PHOLEXSEM treatment were compared to those of a control treatment, i.e., a Promoting Aphasics Communicative Effectiveness (PACE) protocol.

Finally, we studied the effects of age, education, disease duration, brain lesion volume, and functional independence (Functional Idependence Measure, FIM) on the treatment-induced linguistic improvements.

ELIGIBILITY:
Inclusion Criteria:

* acquired brain-damage
* presence of aphasia

Exclusion Criteria:

* global aphasia
* undergoing another treatment for aphasia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Neuropsychological Examination of Language (ENPA) | At baseline and immediately after the intervention.
  A test for aphasia assessment in the Italian population
Change from baseline in phonemic fluency | At baseline and immediately after the intervention.
  To assess lexical retrieval based on a letter
Change from baseline in semantic fluency | At baseline and immediately after the intervention.
  To assess lexical retrieval based on a semantic category
Change from baseline in syntagma repetition | At baseline and immediately after the intervention.
  The syntagma repetition test from the Aachner Aphasie Test (AAT)
Change from baseline in the auditory digit span | At baseline and immediately after the intervention.
  To assess auditory verbal short-term memory
Change from baseline in the word repetition span | At baseline and immediately after the intervention.
  To assess auditory verbal short-term memory, with words stimuli
Change from baseline in the Token Test | At baseline and immediately after the intervention.
  To assess auditory language comprehension

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on Zenodo upon request.